CLINICAL TRIAL: NCT02126423
Title: Prospective Study on Antimicrobial Resistance Rates Following Repeated Courses of Topical Antibiotics for Intravitreal Injection
Brief Title: Resistance to Antibiotics in Patients Receiving Eye Injections
Status: Completed | Type: Observational
Sponsor: Prism Vision Group (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1001
Record Dates: First submitted 2014-04-23; First posted 2014-04-30 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Age-Related Macular Degeneration; Retinal Vein Occlusion; Diabetic Retinopathy
Keywords: Drug Resistance, Microbial
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion; Diabetic Retinopathy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Conjunctival and nasopharyngeal swabs are procured from each patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1st intravitreal injection: Conjunctival and nasopharyngeal swabs are obtained from each treatment-naive patient receiving their 1st intravitreal injection
  Interventions: Other: Conjunctival and nasopharyngeal swabs
- >20 intravitreal injections: Conjunctival and nasopharyngeal swabs are obtained from each patient with >20 intravitreal injection therapies.
  Interventions: Other: Conjunctival and nasopharyngeal swabs

INTERVENTIONS:
Other: Conjunctival and nasopharyngeal swabs — For conjunctival samples, a sterile swab is moistened with ophthalmic balanced salt solution and gently swept along the lower fornix from the medial to the lateral canthi, with all attempts to avoid the eyelashes and eyelids. For nasopharyngeal cultures, the sterile swab is inserted 2 cm into the naris and rotated against the anterior nasal mucosa for 3 seconds.

SUMMARY:
The administration of short courses of topical antibiotic drops before and/or after intravitreal injections is a common practice, but increasing evidence suggests this may not lower the risk of infectious endophthalmitis and could increase rates of antimicrobial resistance. The purpose of the present study is to determine the antimicrobial resistance profiles in patients who have received numerous (≥ 20) courses of antibiotics for intravitreal injection compared with untreated controls.

This study compares 20 control patients without prior intravitreal injection to 20 patients who have undergone ≥ 20 prior intravitreal injections accompanied by a course of topical antibiotics for two days before and/or after the injection procedure. The lower, inner eyelid and nasal cavity were cultured and evaluated via disk diffusion method for antimicrobial sensitivity.

DETAILED DESCRIPTION:
Before administration of anti-VEGF therapy (Vascular Endothelial Growth Factor) or topical antibiotics, conjunctival and nasopharyngeal swabs are procured with the Bacti-Swab transport system (Thermo Fisher Scientific, Waltham, MA). For conjunctival samples, a sterile swab is moistened with ophthalmic balanced salt solution and gently swept along the lower fornix from the medial to the lateral canthi, with all attempts to avoid the eyelashes and eyelids. For nasopharyngeal cultures, the sterile swab is inserted 2 cm into the naris and rotated against the anterior nasal mucosa for 3 seconds.

Culture swabs are then plated onto 5% sheep blood plates and incubated at 37°C for 3 days. Colonies are isolated and identified with API (Analytical Profile Index) Microbial Identification Kits (bioMérieux Inc., Hazelwood, MO). Antibiotic susceptibility is determined using the Kirby Bauer disc diffusion method. Additional data collected includes age, ocular and systemic medical conditions, and the number of intravitreal injections along with anti-VEGF agents used.

Statistical calculations for antibiotic resistance comprises of t-test and and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (above age 18) diagnosed with age-related macular degeneration and receiving their 1st or 20th (or >20th) intravitreal injection therapy.

Exclusion Criteria:

* Those with current use of topical or systemic antibiotics and an active ocular infection or ocular surface disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Kirby Bauer disc diffusion antimicrobial susceptibility | 15 minutes
  One set of conjunctival and nasopharyngeal swabs obtained from patient shortly after recruitment. Antibiotic susceptibility is determined using the Kirby Bauer disc diffusion method for the following antibiotics: amoxicillin/clavulanate, cefazolin, cefoxitin, erythromycin, moxifloxacin, trimethoprim/sulfamethoxazole, linezolid, clindamycin, and doxycycline.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fine, MD, MHSc, Principal Investigator — Prism Vision Group
Locations (1):
- NJ Retina, Edison, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No